CLINICAL TRIAL: NCT02817776
Title: Prospective Review of the Safety and Effectiveness of the THERMOCOOL SMARTTOUCH® SF (STSF) Catheter Evaluated for Treating Symptomatic PersistenT AF (PRECEPT)
Brief Title: Safety and Effectiveness of STSF Catheter Evaluated for Treating Symptomatic Persistent Atrial Fibrillation (PsAF)
Acronym: PRECEPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STSF-159
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
Keywords: Interventional; Radiofrequency Ablation; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment group (Experimental): Pulmonary vein isolation (PVI) by RF ablation treatment with the THERMOCOOL SMARTTOUCH® SF catheter in persistent AF population.
  Interventions: Device: THERMOCOOL SMARTTOUCH® SF catheter

INTERVENTIONS:
Device: THERMOCOOL SMARTTOUCH® SF catheter — Radiofrequency Ablation

SUMMARY:
This is a prospective, multicenter, non-randomized clinical evaluation utilizing the THERMOCOOL SMARTTOUCH® SF catheter compared to a predetermined performance goal.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the safety and effectiveness of the THERMOCOOL SMARTTOUCH® SF catheter in the treatment of drug refractory symptomatic persistent atrial fibrillation (PsAF) following standard electrophysiology mapping and radio frequency (RF) ablation procedures.

ELIGIBILITY:
Inclusion Criteria:

Candidates for this study must meet ALL of the following criteria:

1. Documented symptomatic persistent AF, which is defined as continuous AF sustains beyond 7 days and less than 1 year and is documented by the following:.

   1. Physician's note indicating continuous AF ≥ 7 days but no more than 1 year; AND
   2. Two electrocardiograms (from any forms of rhythm monitoring) showing continuous AF, with electrocardiogram taken at least 7 days apart OR
   3. 24-hour Holter within 90 days of the ablation procedure showing continuous AF
2. Failed at least one antiarrhythmic drug (AAD) (class I or III) as evidenced by recurrent symptomatic AF, or intolerable to the AAD.
3. Age 18 years or older.
4. Signed Patient Informed Consent Form (ICF).
5. Able and willing to comply with all pre-, post-, and follow-up testing and requirements.

Exclusion Criteria:

Candidates for this study will be EXCLUDED from the study if ANY of the following conditions apply:

1. Continuous AF > 12 months (1-Year) (Longstanding Persistent AF)
2. Previous surgical or catheter ablation for atrial fibrillation
3. Any cardiac surgery within the past 2 months (60 days) (includes percutaneous coronary intervention (PCI))
4. Coronary Artery Bypass Graft (CABG) surgery within the past 6 months (180 days)
5. Valvular cardiac surgical/percutaneous procedure (i.e., ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve)
6. Any carotid stenting or endarterectomy
7. Documented left atrial (LA) thrombus on imaging
8. LA size > 50 mm (parasternal long axis view)
9. Left ventricular ejection fraction (LVEF) < 40%
10. Contraindication to anticoagulation (heparin or warfarin)
11. History of blood clotting or bleeding abnormalities
12. MI within the past 2 months (60 days)
13. Documented thromboembolic event (including Transient Ischemic Attack (TIA) within the past 12 months (365 days)
14. Rheumatic Heart Disease
15. Uncontrolled heart failure or New York Heart Association (NYHA) function class III or IV
16. Severe mitral regurgitation (Regurgitant volume ≥ 60 mL/beat, Regurgitant fraction ≥ 50%, and/or Effective regurgitant orifice area ≥ 0.40cm2)
17. Awaiting cardiac transplantation or other cardiac surgery within the next 12 months (365 days)
18. Unstable angina
19. Acute illness or active systemic infection or sepsis
20. AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
21. Diagnosed atrial myxoma.
22. Presence of implanted implantable cardioverter defibrillator (ICD) /cardiac resynchronization therapy defibrillator (CRT-D).
23. Significant pulmonary disease, (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms.
24. Gastroesophageal Reflux Disease (GERD; active requiring significant intervention not including over-the-counter (OTC) medication)
25. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study.
26. Women who are pregnant (as evidenced by pregnancy test if pre-menopausal)
27. Enrollment in an investigational study evaluating another device, biologic, or drug.
28. Presence of intramural thrombus, tumor or other abnormality that precludes vascular access, or manipulation of the catheter.
29. Presence of any other condition that precludes appropriate vascular access.
30. Life expectancy less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Research; Francis Marchlinski, MD, Principal Investigator — University of Pennsylvania; Bruce Koplan, MD, Principal Investigator — Brigham and Women's Hospital; Walid Saliba, MD, Principal Investigator — The Cleveland Clinic; Tristram Banhson, MD, Principal Investigator — Duke University; Scott Pollak, MD, Principal Investigator — AdventHealth; Hugh Calkins, MD, Principal Investigator — Johns Hopkins University; Moussa Mansour, MD, Principal Investigator — Massachusetts General Hospital; Douglas Packer, MD, Principal Investigator — Mayo Clinic Foundation; Srinivas Dukkipati, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Larry Chinitz, MD, Principal Investigator — NYU Langone Medical Center; Saumil Oza, MD, Principal Investigator — St. Vincent's; Anshul Patel, MD, Principal Investigator — Emory University Saint Joseph's Hospital; Robert Fishel, MD, Principal Investigator — JFK Medical Center; William Maddox, MD, Principal Investigator — University of Alabama at Birmingham; Alexander Mazur, MD, Principal Investigator — University of Iowa; Daniel Melby, MD, Principal Investigator — Allina Health System; Christopher Liu, MD, Principal Investigator — New York Presbyterian Hospital; Kenneth Ellenbogen, MD, Principal Investigator — Virginia Commonwealth University; Chad Brodt, MD, Principal Investigator — Stanford University; Laurent Macle, MD, Principal Investigator — Montreal Heart; Philip Gentlesk, MD, Principal Investigator — Sentara Heart Hospital; James B Deville, MD, Principal Investigator — Baylor Research Institute; Charles Athill, MD, Principal Investigator — San Diego Cardiac Center; Craig Delaughter, MD, Principal Investigator — Texas Health Heart & Vascular; Marwan Bahu, MD, Principal Investigator — Phoenix Cardiovascular Research Group; Jose Osorio, MD, Principal Investigator — Affinity Cardiovascular Specialists (Alabama Cardiovascular Group); Marc Deyell, MD, Principal Investigator — St. Paul

REFERENCES:
- [Derived] Natale A, Calkins H, Osorio J, Pollak SJ, Melby D, Marchlinski FE, Athill CA, Delaughter C, Patel AM, Gentlesk PJ, DeVille B, Macle L, Ellenbogen KA, Dukkipati SR, Reddy VY, Mansour M; PRECEPT Investigators. Positive Clinical Benefit on Patient Care, Quality of Life, and Symptoms After Contact Force-Guided Radiofrequency Ablation in Persistent Atrial Fibrillation: Analyses From the PRECEPT Prospective Multicenter Study. Circ Arrhythm Electrophysiol. 2021 Jan;14(1):e008867. doi: 10.1161/CIRCEP.120.008867. Epub 2020 Dec 8. PMID 33290093
- [Derived] Mansour M, Calkins H, Osorio J, Pollak SJ, Melby D, Marchlinski FE, Athill CA, Delaughter C, Patel AM, Gentlesk PJ, DeVille B, Macle L, Ellenbogen KA, Dukkipati SR, Reddy VY, Natale A. Persistent Atrial Fibrillation Ablation With Contact Force-Sensing Catheter: The Prospective Multicenter PRECEPT Trial. JACC Clin Electrophysiol. 2020 Aug;6(8):958-969. doi: 10.1016/j.jacep.2020.04.024. PMID 32819531

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 367 subjects were proposed in the protocol to be enrolled for this study. The enrollment had been completed and closed after reaching a total of 381 enrolled subjects.
  The last subject was enrolled on February 6th, 2018.
Period: Overall Study
Arm/Group | Treatment Group
Started | 381 (33 excluded prior to procedure. 348 had study catheter inserted (Safety Population))
Completed | 293
Not Completed | 88
Not completed — Excluded | 33
Not completed — Lost to Follow-up | 20
Not completed — Withdrawal by Subject | 33
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 381
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.6 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 271
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 357
  Unknown or Not Reported | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 349
  More than one race | 0
  Unknown or Not Reported | 23

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint - Percentage of Participants With Any PAE Within 7 Days
Description: The primary safety endpoint is the incidence of any early onset (within 7 days of the initial and repeat AF ablation procedure) Primary Adverse Events (AE), which are listed below:
  * Death
  * Atrio-esophageal fistula*
  * Cardiac Tamponade**+/Perforation+
  * Myocardial infarction (MI)
  * Stroke / Cerebrovascular accident (CVA) †, ††
  * Thromboembolism
  * Transient Ischemic Attack
  * Diaphragmatic paralysis
  * Pneumothorax
  * Heart block
  * PV stenosis*
  * Pulmonary edema (Respiratory Insufficiency)
  * Pericarditis
  * Major Vascular access complication / bleeding
Time Frame: 7 days (except as noted in analysis population description)
Population: The safety population was used as the primary analysis population. Subjects with missing 3-month follow-up were excluded from the primary analysis unless the subjects experienced a Primary AE prior to the 3-month visit post-procedure. PV stenosis and AE fistula that occurred > 1 week and cardiac tamponade/perforation that occurred up to 30 days post ablation were also deemed Primary AEs.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 344
Percentage of participants | 4.7

2. Primary Outcome: Effectiveness: Freedom From Documented Atrial Fibrillation (AF), Atrial Tachycardia (AT), or Atrial Flutter (AFL) Episodes Through 15-month Follow-up
Description: The primary effectiveness endpoint for this study will be freedom from documented atrial fibrillation (AF), atrial tachycardia (AT), or atrial flutter (AFL) episodes through 15-month follow-up (post 3-Month Medication Adjustment Period followed by a 3-Month Therapy Consolidation period (Day 181-450)) and freedom from the following failure modes:
  * Acute Procedural Failure
  * Non-Study Catheter Failure
  * Repeat Ablation Failure
  * AAD Failure
  * Surgical Failure
Time Frame: 15-month follow-up
Population: The PP population was used as the primary analysis population. Subjects who did not complete the 15-month follow-up were considered missing and were excluded from the primary analysis unless the subjects experienced effectiveness failure prior to exiting the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 297
Percentage of Participants | 59.3

3. Secondary Outcome: Acute Procedural Success
Description: Acute procedural success is defined as confirmation of entrance block in all pulmonary veins.
Time Frame: Immediate post-procedure
Population: Per Protocol Population
Measure: Number; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 333
Participants | 330

4. Secondary Outcome: 15-Month Single Procedure Success
Description: The 15-month single procedure success is defined as freedom from documented AF/AFL/AT recurrence (episodes > 30 secs) during the Evaluation Period after a single ablation procedure. Any repeat ablation procedure during the Evaluation Period will be deemed effectiveness failure for this analysis.
Time Frame: 15-Month
Population: Per Protocol Population, n=333, minus 3 acute procedural failures and 36 missing outcomes not included in primary effectiveness endpoint calculation.
Measure: Number; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 294
Participants | 182

5. Secondary Outcome: Early Onset Serious Adverse Event (SAE)
Description: Occurrence of Early Onset (within 7 days of initial ablation) Serious Adverse Event
Time Frame: 7 days
Population: Safety Population (number of subjects with study catheter inserted) was the analysis population for secondary safety endpoints.
Measure: Number; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 348
Participants | 33

6. Secondary Outcome: Peri-Procedural Serious Adverse Event (SAE)
Description: Peri-Procedural (>7 to 30 days) Serious Adverse Event
Time Frame: >7 to 30 days
Population: Safety Population (number of subjects with study catheter inserted)
Measure: Number; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 348
Participants | 6

7. Secondary Outcome: Late Onset Serious Adverse Event (SAE)
Description: Occurrence of Late Onset (>30 days) Serious Adverse Event
Time Frame: >30 days up to 15 months
Population: Safety Population (number of subjects with study catheter inserted) and excluding subjects who exited prior to 30 days of follow up in the study.
Measure: Number; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 346
Participants | 59

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 2/348
Serious Adverse Events (participants affected / at risk) | 85/348
Other Adverse Events (participants affected / at risk) | 0/348
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=348)
Cardiac Tamponade (Cardiac disorders) | 5 (5)
Cerebrovascular Accident (CVA) / Stroke (Nervous system disorders) | 1 (1)
Diaphragmatic Paralysis (Cardiac disorders) | 1 (1) — Possibly device related and possibly procedure related
Pulmonary Edema (Respiratory Insufficiency) (Cardiac disorders) | 5 (5)
Pericarditis (Cardiac disorders) | 2 (2)
Major Vascular Access Complication / Bleeding (Cardiac disorders) | 3 (3)
Atrial Fribrillation (Cardiac disorders) | 11 (13) — Not Device Related and Not Procedure Related
Atrial Fibrillation (Cardiac disorders) | 1 (1) — Possibly device related
Atrial Fibrillation (Cardiac disorders) | 1 (1) — Possibly procedure related
Esophageal Ulcer (Gastrointestinal disorders) | 1 (1) — Definitely device related
Esophageal Ulcer (Gastrointestinal disorders) | 1 (1) — Definitely procedure related
Bradycardia (Cardiac disorders) | 4 (4) — Not device related
Bradycardia (Cardiac disorders) | 4 (4) — Not procedure related
Chest Pain (Cardiac disorders) | 6 (7) — Not device related
Chest Pain (Cardiac disorders) | 1 (1) — Possibly procedure related
Chest Pain (Cardiac disorders) | 5 (6) — Not procedure related
Complication associated with urinary catheter (General disorders) | 1 (1) — Possibly procedure related, not device related
Complication associated with urinary catheter (General disorders) | 2 (3) — Definitely procedure related, not device related
Diplopia (Eye disorders) | 1 (1) — Not device related
Diplopia (Eye disorders) | 1 (1) — Possibly procedure related
Fluid overload (Metabolism and nutrition disorders) | 2 (2) — Definitely procedure related
Hypertensive Crisis (Vascular disorders) | 1 (1) — Not device related
Hypertensive Crisis (Vascular disorders) | 1 (1) — Not procedure related
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not device related
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Possibly procedure related
Pericardial Effusion (Cardiac disorders) | 2 (2) — Not device related
Pericardial Effusion (Cardiac disorders) | 1 (1) — Possibly procedure related
Pericardial Effusion (Cardiac disorders) | 1 (1) — Not procedure related
Pyrexia (General disorders) | 1 (1) — Not device related
Pyrexia (General disorders) | 1 (1) — Not procedure related
Renal Failure (Renal and urinary disorders) | 1 (1) — Not device related
Renal Failure (Renal and urinary disorders) | 1 (1) — Possibly procedure related
Sepsis (Infections and infestations) | 3 (3) — Not device related
Sepsis (Infections and infestations) | 1 (1) — Definitely procedure related
Sepsis (Infections and infestations) | 2 (2) — Not procedure related
Tachycardia (Cardiac disorders) | 11 (11) — Not device related
Tachycardia (Cardiac disorders) | 10 (10) — Not procedure related
Tachycardia (Cardiac disorders) | 1 (1) — Possibly procedure related
Torsade de pointes (Cardiac disorders) | 1 (1) — Not device related
Torsade de pointes (Cardiac disorders) | 1 (1) — Not procedure related
Urinary tract infection (Renal and urinary disorders) | 1 (1) — Not device related
Urinary tract infection (Renal and urinary disorders) | 1 (1) — Possibly procedure related
Atrial flutter (Cardiac disorders) | 6 (7) — Not device related
Atrial flutter (Cardiac disorders) | 5 (5) — Not procedure related
Atrial flutter (Cardiac disorders) | 1 (1) — Possibly device related
Atrial flutter (Cardiac disorders) | 1 (1) — Definitely procedure related
Atrial flutter (Cardiac disorders) | 2 (2) — possibly procedure related
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Not device related
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Possibly procedure related
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not procedure related
Presyncope (Nervous system disorders) | 1 (1) — Not device related
Presyncope (Nervous system disorders) | 1 (1) — Not procedure related
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Not device related
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Possibly procedure related
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not procedure related
Tuberculosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not procedure related
Tuberculosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not device related
Abdominal pain (Gastrointestinal disorders) | 1 (1) — Not device related
Abdominal pain (Gastrointestinal disorders) | 1 (1) — Not procedure related
Arrhythmia (Cardiac disorders) | 2 (2) — Not device related
Arrhythmia (Cardiac disorders) | 1 (1) — Possibly procedure related
Arrhythmia (Cardiac disorders) | 1 (1) — Not procedure related
Atrioventricular block (Cardiac disorders) | 1 (1) — Not device related
Atrioventricular block (Cardiac disorders) | 1 (1) — Not procedure related
Back disorder (Musculoskeletal and connective tissue disorders) | 1 (1) — Not device related
Back disorder (Musculoskeletal and connective tissue disorders) | 1 (1) — Not procedure related
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Not device related
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Not procedure related
Bronchitis viral (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not device related
Bronchitis viral (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not procedure related
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) — Not device related
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) — Not procedure related
Cardiac Failure (Cardiac disorders) | 1 (1) — Not device related
Cardiac Failure (Cardiac disorders) | 1 (1) — Not procedure related
Cardiac failure congestive (Cardiac disorders) | 4 (4) — Not device related
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) — Possibly procedure related
Cardiac Failure Congestive (Cardiac disorders) | 3 (3) — Not procedure related
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) — Not device related
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) — Not procedure related
Cholecystitis (Hepatobiliary disorders) | 1 (1) — Not device related
Cholecystitis (Hepatobiliary disorders) | 1 (1) — Not procedure related
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not device related
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not procedure related
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not device related
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not procedure related
Coronary artery occlusion (Cardiac disorders) | 1 (1) — Not device related
Coronary artery occlusion (Cardiac disorders) | 1 (1) — Not procedure related
Device related infection (Infections and infestations) | 1 (1) — Not device related
Device related infection (Infections and infestations) | 1 (1) — Not procedure related
Femur Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Not device related
Hematuria (Renal and urinary disorders) | 1 (1) — Not device related
Hematuria (Renal and urinary disorders) | 1 (1) — Not procedure related
Hemorrhage (Vascular disorders) | 2 (2) — Not device related
Hemorrhage (Vascular disorders) | 2 (2) — Not procedure related
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Not device related
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Not procedure related
Hypersensitivity (Immune system disorders) | 1 (1) — Not device related
Hypersensitivity (Immune system disorders) | 1 (1) — Not procedure related
Influenza (Infections and infestations) | 2 (2) — Not device related
Influenza (Infections and infestations) | 2 (2) — Not procedure related
Intra-abdominal hematoma (Gastrointestinal disorders) | 1 (1) — Not device related
Intra-abdominal hematoma (Gastrointestinal disorders) | 1 (1) — Not procedure related
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not device related
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not procedure related
Major depression (Psychiatric disorders) | 1 (1) — Not device related
Major depression (Psychiatric disorders) | 1 (1) — Not procedure related
Myocardial infarction (Cardiac disorders) | 2 (2) — Not device related
Myocardial infarction (Cardiac disorders) | 2 (2) — Not procedure related
Obesity (Metabolism and nutrition disorders) | 1 (1) — Not device related
Obesity (Metabolism and nutrition disorders) | 1 (1) — Not procedure related
Esophageal stenosis (Gastrointestinal disorders) | 1 (1) — Not device related
Esophageal stenosis (Gastrointestinal disorders) | 1 (1) — Not procedure related
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) — Not device related
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) — Not procedure related
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Not device related
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Not procedure related
Pneumonia (Infections and infestations) | 3 (3) — Not device related
Pneumonia (Infections and infestations) | 3 (3) — Not procedure related
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Not device related
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Not procedure related
Seroma (Injury, poisoning and procedural complications) | 1 (1) — Not device related
Seroma (Injury, poisoning and procedural complications) | 1 (1) — Not procedure related
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) — Not device related
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) — Not procedure related
Squamous cell cercinoma (Skin and subcutaneous tissue disorders) | 1 (1) — Not device related
Squamous cell cercinoma (Skin and subcutaneous tissue disorders) | 1 (1) — Not procedure related
Syncope (Nervous system disorders) | 1 (1) — Not device related
Syncope (Nervous system disorders) | 1 (1) — Not procedure related
Tremor (Nervous system disorders) | 1 (1) — Not device related
Tremor (Nervous system disorders) | 1 (1) — Not procedure related
Ventricular extrasystoles (Cardiac disorders) | 1 (1) — Not device related
Ventricular extrasystoles (Cardiac disorders) | 1 (1) — Not procedure related
Vertigo (Ear and labyrinth disorders) | 1 (1) — Not device related
Vertigo (Ear and labyrinth disorders) | 1 (1) — Not procedure related
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Not device related
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Possibly procedure related
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not procedure related
Fluid Overload (Metabolism and nutrition disorders) | 2 (2) — Not device related
Cerebrovascular accident (CVA) / Stroke (Nervous system disorders) | 1 (1) — Not procedure or device related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/76/NCT02817776/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT02817776/SAP_001.pdf